CLINICAL TRIAL: NCT07180693
Title: Breast Cancer RElapsed in Patients Treated With Adjuvant CDK4/6 Inhibitors: Evaluation in the Real-world Setting
Brief Title: Breast Cancer RElapsed in Patients Treated With Adjuvant CDK4/6 Inhibitors:
Acronym: BREAKER
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: UID 4879
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Adjuvant Therapy; CDK4/6 Inhibitor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Patients undergoing treatment with CDK4/6 inhibitors

SUMMARY:
This is a multicenter observational study with both retrospective and prospective phase, designed to evaluate the clinico-pathologic characteristics and outcomes of patients with HR+/HER2- EBC at high risk of recurrence treated with ribociclib or abemaciclib in combination with ET in the adjuvant setting.

DETAILED DESCRIPTION:
The study will also evaluate clinico-pathologic characteristics, patterns of recurrence, therapeutic choices and outcomes of the subgroup of patients relapsed during or within 12 months after adjuvant therapy with CDK4/6 inhibitors in combination with ET.

ELIGIBILITY:
Inclusion Criteria:

* Female (regardless of menopausal status) or male ≥18 years of age;
* The patient has confirmed HR+, HER2-, early-stage resected invasive breast cancer candidate to adjuvant CDK4/6 inhibitors (abemaciclib or ribociclib);
* ER and PgR positivity is defined as evidence of immunohistochemical staining ≥ 1% according to ASCO/CAP recommendations; HER2 negativity is defined as expression of the membrane protein in immunohistochemistry 0 or 1+ or with a 2+ in situ hybridization (ISH) test negative as per ASCO/CAP recommendations;
* Patients who are initiating or have initiated adjuvant treatment with a CDK4/6 inhibitor (abemaciclib or ribociclib) in combination with endocrine therapy (ET). Treatment must have started on or after January 1, 2021.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
* Consent to data treatment according to the local regulation.

Exclusion Criteria:

* Current participation in any other HR+/HER2- EBC study with any investigational products;
* Patients who have already received adjuvant treatment with a CDK4/6 inhibitor as part of a clinical trial;
* Patients unable to comply with the requirements of the study or who, in the judge of the study physician, should not be included in the study;
* Patients with a history of previous BC, with the exception of Ductal carcinoma in situ (DCIS) treated by locoregional therapy alone ≥5 years ago;
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission with no therapy for a minimum of 5 years from the index date, will be excluded, as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with HR+/HER2- breast cancer who have received medical treatment in the neoadjuvant or adjuvant setting (chemotherapy, radiotherapy and hormonotherapy) and who have received or are scheduled to initiate adjuvant treatment with CDK4/6 inhibitors (abemaciclib or ribociclib) in combination with ET in the adjuvant setting.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2030-08-01 (Estimated)

PRIMARY OUTCOMES:
Invasive-disease free survival (IDFS) | 3 years
  Invasive disease-free survival (IDFS) will be defined as the time from surgery to invasive loco-regional recurrence, metastasis, other primary non-breast carcinomas, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Distant relapse-free survival (DRFS) | 5 years
  DRFS will be defined as the time from surgery to distant recurrence or death from any cause, whichever occurs first.
progression-free survival (PFS) | 5 years
  PFS will be defined as the time from the disease recurrence to the date of documented disease progression or death from any cause, whichever occurs first.
Overall survival (OS) | 5 years
  OS will be defined as the time from surgery to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Bianco, MD, Study Chair — European Institute of Oncology
Locations (18):
- Italy (18):
  - ASST Papa Giovanni XXIII, Bergamo, Italy
  - ASST Spedali Civili di Brescia, Brescia, Italy
  - P.O. Antonio Perrino - ASL Brindisi, Brindisi, Italy
  - ASST Ospedale Maggiore di Crema, Crema, Italy
  - ASST Lecco - PO Alessandro Manzoni, Lecco, Italy
  - Asst Ovest Milanese, Legnano, Italy
  - IRCCS Ospedale San Raffaele, Milan, Italy
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan, Italy
  - European Institute of Oncology, Milan, Italy
  - PO Luigi Sacco - ASST Fatebenefratelli Sacco, Milan, Italy
  - Azienda Ospedaliero-Universitaria di Modena, Modena, Italy
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Italy
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli, Italy
  - ICS Maugeri IRCCS, Pavia, Italy
  - Policlinico San Matteo, Pavia, Italy
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, Italy
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italy
  - Ospedale Isola Tiberina - Gemelli Isola, Roma, Italy